CLINICAL TRIAL: NCT02663596
Title: A Prospective, Open-Label Study of the Safety and Therapeutic Drug Monitoring of Continuous Infusion Vancomycin Through the Addition of the Vancomycin Into the Continuous Renal Replacement Therapy Solution
Brief Title: Safety and TDM of Continuous Infusion Vancomycin Through Continuous Renal Replacement Therapy Solution
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Drexel University (Other)
Collaborators: The Center for Pediatric Pharmacotherapy, LLC (Unknown)
Responsible Party: Principal Investigator, Jeffrey J. Cies,PharmD,MPH,BCPS-AQ ID,BCPPS,FCCP,FCCM,FPPAG, Pharmacy Clinical Coordinator, Critical Care and Infectious Diseases Clinical Pharmacist, Drexel University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol 1510004004
Record Dates: First submitted 2016-01-12; First posted 2016-01-26 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Pediatric Continuous Renal Replacement Therapy; Dialysis; Renal Failure
Keywords: Pediatric; Continuous Renal Replacement Therapy; Dialysis; Therapeutic drug monitoring; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Renal Insufficiency | interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vancomycin (Experimental): Patients with vancomycin mixed in the CRRT solution(s)
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Vancomycin — Patient requiring CRRT and vancomycin that provide consent will be given vancomycin as a continuous infusion by mixing the vancomycin into the CRRT solution(s)
  Other Names: Continuous renal replacement therapy solutions

SUMMARY:
The purpose of this investigation is to evaluate the safety of delivering continuous infusion (CI) vancomycin in pediatric CRRT by utilizing CI via by mixing the vancomycin into the CRRT solution(s). The secondary objectives are to describe the ability to achieve therapeutic vancomycin concentrations by utilizing this new delivery technique.

Primary Objectives:

To determine whether delivering continuous infusion vancomycin mixed into the CRRT solution can maintain therapeutic levels of drug in patients being treated for proven or suspected Gram-positive bacterial infections.

DETAILED DESCRIPTION:
Treatment Patients deemed candidates for CRRT and antimicrobial therapy for a proven or suspected Gram-positive bacterial infection that includes vancomycin at the time of CRRT initiation or at any time during the CRRT course. If vancomycin is part of the empiric regimen or needed for definitive therapy an assessment will be made whether the vancomycin can be administered via a continuous infusion by mixing the vancomycin in the CRRT solution(s).

Intervention Administration of continuous infusion vancomycin via mixing vancomycin in the CRRT solution(s). The CRRT solution will be prepared at the time it is needed following current standard operating procedures of the Department of Pharmacy at St. Christopher's Hospital for Children for sterile product compounding. The amount of vancomycin to be added to the CRRT solution will be determined by the clinical condition such as the site of infection,infecting organism(s), and serum drug levels. The mixed solution will be infused for the duration it is prescribed for CRRT. Vancomycin is stable with the components of the CRRT solution for at least 96 hours, therefore the frequency with which each CRRT solution bag will be prepared will not exceed 96 hours.

Vancomycin dosing and concentration adjustments:

For patients started on vancomycin after initiation of CRRT, a single loading dose of 15-20 mg/kg of total body weight will be given intravenously over 60 minutes, after which the vancomycin will be added directly to the CRRT solution(s). Vancomycin will be added at a final concentration of 30 mg/L at CRRT initiation, regardless of age. For patients receiving vancomycin prior to the initiation of CRRT, if the last dose administered is > 8 hours prior to CRRT initiation, a loading dose of 15-20 mg/kg of total body weight will be given intravenously over 60 minutes, after which the vancomycin will be added directly to the CRRT solution(s). Vancomycin will be added at a final concentration of 30 mg/L at CRRT initiation, regardless of age. The first serum vancomycin level will be determined 8-12 hours after initiation of CRRT mixed with vancomycin. All serum for vancomycin concentrations determination will be obtained directly from the patient via a central line, arterial line or peripheral venipuncture and no vancomycin concentrations will obtained from the CRRT circuit for analysis.

Vancomycin concentrations in the CRRT solution(s) will be adjusted based on the initial vancomycin serum plateau level, and subsequent levels will be obtained based on these changes. The target vancomycin plateau serum concentrations range is 15-30 mg/L. If the first vancomycin plateau level obtained is within range, daily vancomycin plateau levels will be obtained for the duration the vancomycin is mixed in the CRRT solution. If the first vancomycin plateau level is not within range, the vancomycin concentration in the CRRT solution will be adjusted. Subsequent vancomycin plateau levels will be obtained 8-12 hours after the vancomycin concentration change and this process will continue until a therapeutic plateau level is obtained. Once a therapeutic plateau level is obtained, daily vancomycin plateau levels will be obtained for the duration the vancomycin is mixed in the CRRT solution.

Blood samples for vancomycin analysis will be obtained 8-12 hours after starting the CRRT solution mixed with vancomycin. Based on the first drug level obtained, changes to the concentration may be made to adjust to the desired serum concentration and serum levels will be obtained 8-12 hours after each change to the vancomycin concentration in the CRRT solution. Once a therapeutic level is obtained, serum levels will be obtained as needed but usually not more frequently than daily.

If the first vancomycin plateau level is < 10 mcg/mL, then a single, supplemental dose of 10 mg/kg of vancomycin will be given while the vancomycin CRRT concentration is being adjusted.

ELIGIBILITY:
Inclusion Criteria

Patients eligible to participate in the study must meet all of the following criteria prior to any study-related procedure:

1. The need for continuous renal replacement therapy (CRRT) of any modality

1. CVVH-continuous veno-venous hemofiltration
2. CVVHD-continuous veno-venous hemodialysis
3. CVVHDF-continuous veno-venous hemodiafiltration

2. Documented or suspected Gram-positive bacterial infection necessitating the use of vancomycin while receiving CRRT.

Exclusion Criteria

Patients will be considered ineligible if they meet any of the following criteria:

1. History of any moderate or severe hypersensitivity or allergic reaction to vancomcyin (a history of mild rash followed by uneventful re-exposure and/or red man syndrome is not a contraindication)
2. Any rapidly-progressing disease or immediately life-threatening illness (defined as imminent death within 48 hours in the opinion of the investigator)
3. Any condition or circumstance that, in the opinion of the investigator, would compromise the safety of the patient or the quality of study data
4. Planned or prior participation in any other interventional drug study within 30 days
5. Females that are pregnant or breastfeeding

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with therapeutic vancomycin serum levels | Until the end of the study, up to 33 months
  The CRRT circuit (tubing, filter) will be inspected and evaluated for flow rates and clotting hourly

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J Cies, PharmD, MPH, Principal Investigator — Drexel University
Locations (1):
- St. Christopher's Hospital for Children, Philadelphia, Pennsylvania, United States